CLINICAL TRIAL: NCT07365566
Title: Pain Assessment in Patients With Idiopathic REM Sleep Behaviour Disorder
Acronym: PAIN-iRBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/25/0567; ID-RCB (Other: 2025-A02575-44)
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: REM Sleep Behavior Disorder (iRBD); Narcolepsy Type 1
Keywords: parkinson; REM sleep; pain; REM sleep behavior disorder; narcolepsy Type 1; sleep
MeSH Terms: conditions — REM Sleep Behavior Disorder; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idiopathic REM sleep Behavior disorder (iRBD) Group (Experimental): Patients who have an idiopathic REM sleep Behavior Disorder
  Interventions: Other: Thermo test pain; Other: Pain questionnaires; Other: No motors symptoms evaluations
- Idiopathic REM Sleep Bhavior Disorder (iRBD) + narcolepsy type 1 (Active Comparator): patients who have an iRBD and who have type 1 narcolepsy
  Interventions: Other: Thermo test pain; Other: Pain questionnaires; Other: No motors symptoms evaluations

INTERVENTIONS:
Other: Thermo test pain — Patients will undergo a pain test, also called a thermotest, which consists of determining pain thresholds using a thermometer applied to the hand.
Other: Pain questionnaires — Patients will complete various questionnaires about pain
Other: No motors symptoms evaluations — Patients will complete questionnaires

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder after Alzheimer's disease, with over 12 million patients expected globally by 2040. The disease is currently diagnosed at the appearance of motor symptoms, but by then, over 60% of striatal dopaminergic neurons have already been destroyed. Prodromal symptoms such as idiopathic REM Sleep Behavior Disorder (iRBD), anosmia, mood disorders and constipation appear earlier and are listed as criteria for a prodromal PD diagnosis. Identifying early signs is critical to initiate neuroprotective treatments as early as possible. While pain is prevalent and highly disabling in early PD, no data are currently available on pain perception in iRBD patients, whose condition is of the main risk factor for PD development.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with iRBD confirmed by polysomnography;
* No clinical diagnosis of Parkinson's disease or other diagnosis of neurodegenerative disease;
* Ability to understand and complete study procedures and questionnaires;

Control group:

* Diagnosed with narcolepsy type 1;
* Coexisting REM sleep behavior disorder confirmed by polysomnography;
* Ability to understand and complete study procedures and questionnaires;

Exclusion Criteria:

* Diagnosed Parkinson's Disease, dementia with Lewy bodies or multiple system atrophy;
* Severe depression according to Diagnostic and Statistical Manual of Mental Disorders (DSM V);
* Inability to complete study procedures or questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the intensity of chronic pain between patients with iRBD and a control group of patients | 2 hours after the inclusion
  Measuring the Visual Analog Scale (VAS) between patients with iRBD without diagnosis of PD and a control group of patients diagnosed with narcolepsy type 1 who present RBD (Rapid eye movement sleep behavior disorder).

SECONDARY OUTCOMES:
Describe semiological characteristics of pain in RBD patients | 2 hours after the inclusion
  Description of characteristics of pain
Compare the presence of chronic pain | 2 hours after the inclusion
  Number of patients with chronic pain in both groups for at least 3 months.
Assessing Pain Characteristics | 2 hours after the inclusion
  Score obtained on pain questionnaires
Assessment of thermal pain threshold and tolerance | 2 hours after the inclusion
  Results of the quantitative sensory test (thermal thermotest) in both groups
Assessment of correlations between the intensity of chronic pain | 2 hours after the inclusion
  Correlation between Visual Analogue Scale (VAS) measurements and questionnaire responses

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Expert Parkinson Hôpital Pierre Paul Riquet Place du Docteur Baylac, Toulouse, France

IPD SHARING:
Plan to Share IPD: No